CLINICAL TRIAL: NCT04978246
Title: Evaluation Of Cognitive Functions In Adult Individuals With COVID-19
Brief Title: Cognitive Functions After COVID-19
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Büşra Tüfekçi, Principal Investigator, Medipol University
Other Study IDs: Medipol Mega3
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Cognitive Decline
Keywords: Cognitive Functions; COVID-19; Attention; Executive Functions; Memory; Neurophysiology
MeSH Terms: conditions — Cognitive Dysfunction; COVID-19 | interventions — Stroop Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The study group consists of 50 individuals aged 18-50 years who have received a positive COVID-19 RT-PCR test in the past 60 days.
  Interventions: Behavioral: Neuropsychometric Test
- Control Group: The control group consists of 50 healthy individuals aged 18-50 years who have not had COVID-19.
  Interventions: Behavioral: Neuropsychometric Test

INTERVENTIONS:
Behavioral: Neuropsychometric Test — Participants' global cognitive skills were measured by the Montreal Cognitive Assessment Test (MoCA), the Clock Drawing Test and memory functions, the Öktem Verbal Memory Processes Test (Ö-SBST), the attention functions by the Digit Span Forward and Digit Span Backwards Test, the executive functions by Categorical Fluency, Phonemic Fluency, the Stroop Test, Trail Making Test A and B, visuospatial skills were evaluated with the Rey-Osterrieth Complex Figure Test (ROCF), and behavioral symptoms were evaluated with the Neuropsychiatric Inventory (NPI).
  Other Names: Montreal Cognitive Assessment Test (MoCA); Clock Drawing Test; Öktem Verbal Memory Processes Test (Ö-SBST); Digit Span Forward Test; Digit Span Backwards Test; Categorical Fluency; Phonemic Fluency; Stroop Test; Trail Making Test A; Trail Making Test B; Rey-Osterrieth Complex Figure Test (ROCF); Neuropsychiatric Inventory (NPI)

SUMMARY:
This study was aimed to evaluate the post-infection cognitive functions of adult individuals with COVID-19. 50 individuals with COVID-19 and 50 healthy control groups were included in the study. Cognitive functions of individuals with COVID19 compared with healthy individuals.

DETAILED DESCRIPTION:
This study was aimed to evaluate the post-infection cognitive functions of adult individuals with COVID-19. Fifty COVID-19 patients, aged between 18-50 years, who had positive RT-PCR test in the last 60 days and later recovered, were included in the study. The study group was compared with the control group consisting of 50 healthy individuals in whom gender, age and education year has not difference significantly. Participants' global cognitive skills were measured by the Montreal Cognitive Assessment Test (MoCA), the Clock Drawing Test and memory functions, the Öktem Verbal Memory Processes Test (Ö-SBST), the attention functions by the Digit Span Forward and Digit Span Backwards Test, the executive functions by Categorical Fluency, Phonemic Fluency, the Stroop Test, Trail Making Test A and B, visuospatial skills were evaluated with the Rey-Osterrieth Complex Figure Test (ROCF), and behavioral symptoms were evaluated with the Neuropsychiatric Inventory (NPI). The study group was evaluated between 21 and 60 days from the onset of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Having positive for the COVID-19 RT-PCR test and turned negative in the last 60 days.
* be 18-50 years old
* 21 days have passed since the onset of the disease

Exclusion Criteria:

* Having any neurological or psychiatric illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Test (MoCA) | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  It is a test that measures attention and concentration, executive functions, memory, language, visuospatial skills, abstract thinking, calculation and orientation skills in order to distinguish individuals with mild cognitive impairment from healthy individuals.

SECONDARY OUTCOMES:
Clock Drawing Test | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The person is asked to draw a clock circle and place numbers in it. After succeeding, they are asked to show 11 by 10 crossing. This test can test comprehension, memory, visuospatial functions and executive functions.
Öktem Verbal Memory Processes Test (Ö-SBST) | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The test consists of fifteen unrelated words. Fifteen words are read to the subject at one-second intervals and then asked to say the ones that come to mind. In this process, information is collected about the subject's ability to maintain instant memory and attention. The number of correct answers of the subject is recorded as Instant Memory Score. After the first attempt, the same list is read to the subject nine more times, and each time he is asked to say all he remembers. This gives information about the subject's learning ability.
Digit Span | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The test consists of two parts as forward and backward span. In the forward digit span, the numbers are read at one second intervals and the patient is asked to repeat the randomly read numbers in the same order. It assesses attention and short-term memory. In the back digit span, it is requested to repeat the numbers read from the end to the beginning. Working memory is evaluated in the back count range. As the person succeeds in the trials, the test is continued by increasing one step. If the patient fails twice in a row for both sections, the test is discontinued.
Verbal Fluency Test | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  Verbal fluency tests aim to evaluate the executive aspects of verbal behavior by using language capacity as a fluent speech. Verbal fluency tests are applied in two ways: phonemic fluency and semantic fluency. In the semantic fluency test, the person is asked to count animal names in one minute, and in the phonemic fluency test, the person is asked to produce words that start with a certain letter (K-A-S) and are not proper nouns.
Stroop Test | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The Stroop test evaluates focused attention, the ability to change attention in line with changing demands and under a distraction, the ability to suppress a habitual behavior pattern and perform an unusual behavior.
Trail Making Test | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The trail making test consists of two parts, A and B. In part A, the participants are asked to combine the circles with the numbers in the correct order and following each other (1-2-3-4-5...). In section B, there are letters and numbers placed in circles. Participants are asked to combine letters and numbers in the correct sequence (1-A-2-B-3-C-4-D...). The times of both sections are recorded. The A part of the IST evaluates the processing speed based on visual scanning ability, and the B part evaluates the complex attention, planning, set changing, blocking ability and following the sequentiality.
Rey-Osterrieth Complex Figure Test (ROCF) | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The purpose of the test is to evaluate visuospatial structuring skills and visual memory. The test material consists of a complex shape printed on a card, a registration form, an identification form with 24 details, three blank sheets of paper, a pencil and an eraser. The subject is first asked to copy the complex shape and the copying time is noted. During copying, the subject is not informed that he will draw the shape again. In the next step, the complex shape is removed and the person is asked to draw the shape again as far as he can remember, and the drawing time is noted. This is instant recall application. After the instant recall, the subject is not informed that he will draw the shape again, and the subject's mind is occupied by introducing different tests. After 30 minutes, he is asked to draw again. This is the delayed recall phase.
Neuropsychiatric Inventory (NPI) | Any day between 21-60 days from the date of COVID-10 RT-PCR test positive.
  The scale is scored by interview with the patient's relative. A total of 12 behavioral domains (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy, disinhibition, irritability/lability, abnormal motor behavior, sleep/night behaviors, appetite and eating changes) are questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Tüfekçi, MD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Beykoz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Zhou H, Lu S, Chen J, Wei N, Wang D, Lyu H, Shi C, Hu S. The landscape of cognitive function in recovered COVID-19 patients. J Psychiatr Res. 2020 Oct;129:98-102. doi: 10.1016/j.jpsychires.2020.06.022. Epub 2020 Jun 30. PMID 32912598